CLINICAL TRIAL: NCT03175718
Title: The Effect of INPWT on Wound Complications and Clinical Outcomes Following Lower Extremity Sarcoma Surgery in Patients Treated With Preoperative Radiation Therapy: A Multicentre Randomized Controlled Trial
Brief Title: INPWT on Wound Complications & Clinical Outcomes After Lower Extremity Sarcoma Surgery Preop Radiation Therapy Patients
Acronym: VAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. J. Werier (Other)
Responsible Party: Sponsor-Investigator, Dr. J. Werier, Orthopedic Oncologist Surgeon, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170154
Record Dates: First submitted 2017-03-01; First posted 2017-06-05 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Soft-tissue Sarcoma; Wound Complication
Keywords: Sarcoma; Wound; Therapy
MeSH Terms: conditions — Sarcoma; Wounds and Injuries | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: This is a Canadian multicenter superiority randomized clinical trial in patients who are scheduled to undergo surgical resection of a soft tissue sarcoma treated with either preoperative or postoperative radiation therapy and a primary closure. The participants are randomized to Incisional Negative Pressure Wound Therapy (Acelity) or conventional gauze dressing; the current standard of care.
Who Masked: Participant, Outcomes Assessor
Masking Description: The operative team will remain blinded to the dressing until the time of application. Since wound failure requires the need of medical or surgical intervention, primary outcome of this study is not blinded. However, the treatment arm will be blinded to the Research Coordinator/Outcomes Assessor of secondary outcomes including scar assessment, QoL and Functional Assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAC Wound Dressing (Experimental): Limb salvage surgery is performed on sarcoma patients 4-6 week post radiotherapy. These patients will be randomized to receive 7 days of Incisional Negative pressure wound therapy.
  Interventions: Other: Incisional Negative Pressure Wound Therapy (INPWT)
- Control Wound Dressing (Active Comparator): Limb salvage surgery is performed on sarcoma patients 4-6 week post radiotherapy. These patients will be randomized to receive standard gauze dressing with no negative pressure application.
  Interventions: Other: Wound Dressing

INTERVENTIONS:
Other: Incisional Negative Pressure Wound Therapy (INPWT) — A total of 291 patients will be randomized to receive 7 days of Incisional Negative pressure wound dressing. The dressing will be removed 1 week after surgery.
  Arms: VAC Wound Dressing
Other: Wound Dressing — A total of 291 patients will be randomized for standard gauze dressing. This dressing requires no pressure and is applied according to the current standard dressing procedures of the institution. The dressing will be changed every 2-3 days.
  Arms: Control Wound Dressing

SUMMARY:
Project Summary - Aggressive soft tissue cancers are commonly treated with radiation followed by surgery. These wounds have a very high rate of wound complications and infection (30%), resulting in more surgeries, longer hospital stays and complex nursing care. Previous research shows that negative pressure (vacuum) dressings applied to the incision at the end of surgery can reduce these complications. The Investigator and his team across Canada will perform a clinical trial comparing standard dressings to these vacuum dressings. The results of this study have the potential to immediately improve the quality of life of soft tissue cancer patients. It can also decrease the amount of time required in hospital and reduce the cost to the Canadian healthcare system.

DETAILED DESCRIPTION:
This is a multi-center randomized clinical trial lead by the Investigator from the Ottawa Hospital and six other orthopedic cancer centers. The Investigator and the team will be recruiting 248 patients diagnosed with soft tissue cancer who will be treated with radiation therapy followed by surgery. Each of these patients will be randomly assigned to receiving either 7 days of vacuum dressing (Incisional Negative Pressure Wound Therapy) or a standard dressing. Besides this, patients will receive as identical care as possible. The team will then closely follow these patients over a period of 4 month to examine differences in wound complications, length of hospital stay, patient quality of life, patient satisfaction and function. Statistical analysis will be completed by The Ottawa Methods Center and ethical approval will be obtained at each participating site.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older and are able to provide written consent.
* Patients with lower extremity soft tissue sarcoma confirmed by tissue pathology.Each patient must have local cross sectional imaging (CT or MRI) and a staging CT chest.
* Patients eligible for treatment with preoperative radiation therapy followed by limb salvage surgery.
* Patients for which a primary closure must be attained at the time of surgery.
* Patient must be available for postoperative follow-up at the treating center.

Exclusion Criteria:

* Patients who are less than 18 years of age.
* Patients with a benign disease or with prior radiation to the anatomic region in the remote past (not associated with current treatment radiation plans).
* Patients who underwent surgical amputation
* Patients in which primary closure was not achieved (including free flaps and split thickness skin grafts).
* Patients with a life expectancy less than 120 days.
* Patients who have an allergy or sensitivity to adhesive dressings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Wound Complication including re-operation for superficial or deep site infection | 120 days post op
  * Wound requiring deep wound packing to an area greater than 2cm in length
  * Wound requiring persistent dressing changes for greater than 6 weeks. Wound packing and persistent requirement to change the dressing will reflect if the patient has a wound complication.

SECONDARY OUTCOMES:
patient satisfaction | All within this 120 day post-op
  Patient satisfaction will be evaluated by validated questionnaires.
Functional outcome | 120 days postop
  Secondary outcomes include length of stay in hospital,
Overall cost | 120 days
  A cost analysis will be performed by evaluating the average inpatient cost per day, number of emergency department and clinic visits, cost of secondary procedures cost of INPWT and cost of home care visits.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Werier, Principal Investigator — Surgeon
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No